CLINICAL TRIAL: NCT04163965
Title: Data Collection for Pacemaker Recognition Through Capacitive ECG
Acronym: HSM-cECG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Nikolaus Marx, Univ.-Prof. Dr. med., RWTH Aachen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-104
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Pacemaker DDD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients having a pacemaker (Other): Patients having a pacemaker will sit down on a seat bearing capacitive ECG electrodes during their routine heart checkup at the cardiology. Simultaneously standard routine ECG measurements will take place.
  Interventions: Device: Capacitive ECG

INTERVENTIONS:
Device: Capacitive ECG — Patients having a pacemaker will sit down on a seat bearing capacitive ECG electrodes during their routine heart checkup at the cardiology.

SUMMARY:
This study evaluates the signal quality of capacitive ECG (cECG) on pacemaker patients and whether paced rhythms of the pacemaker can be distinguished from the normal beats using cECG signals.

DETAILED DESCRIPTION:
In contrast to classical gold-standard ECG, cECG electrodes can sense the electrical activity of the heart even over the clothing of the subject, which allows several applications in out-of-hospital monitoring. The proposed scenarios for cECG revolve around the unobtrusiveness of the measurement with an inferior signal quality to gold standard ECG. The electrical spikes, that come into existence due to the paced rhythms given by a pacemaker, are only visible in ECG signals recorded by adequate medical instrumentation. Whether cECG can deliver enough signal quality to identify the electrical spikes of the paced rhythms needs to be investigated by recording simultaneous normal and capacitive ECG signals.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an implanted pacemaker
* Subject is under ambulatory or stationary treatment in Uniklinik RWTH Aachen
* Subject gives his/her written consent
* Subject is legally and mentally competent to follow the instructions

Exclusion Criteria:

* Subject has other electrically active implants
* Cardiopulmonary or hemodynamically unstable subjects
* Subject is placed in a judicial institution
* Subject is in a dependency or employment relationship with the examiner
* Subject is legally or mentally unable to give consent for the participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Paced Rhythm Identification | up to 10 weeks after the data collection is completed for each patient
  Cardiologists are asked to classify the heart-beats as "paced" and "normal" in a blind test of mixed normal and capacitive ECG recordings.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No